CLINICAL TRIAL: NCT04033783
Title: The Impact of Walking Behind the Patient on Six-Minute Walk Test Distance in Chronic Obstructive Pulmonary Disease: a Randomized Cross-over Study
Brief Title: Impact of Walking Behind the COPD Patient on 6MWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-00827
Record Dates: First submitted 2019-07-08; First posted 2019-07-26 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: COPD
Keywords: Six minute walk test; Field test; Exercise capacity; Functional capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6MWT - assessor walks behind the patient (Experimental): In this experimental condition, the assessor walks behind the patient to continuously measure oxygen saturation during the test (recommended procedure)
  Interventions: Other: 6MWT - accompanied
- 6MWT - assessor does not walk behind the patient (Active Comparator): In this experimental condition, the assessor does not walk behind the patient. The patient carries the pulse oximeter to continuously measure oxygen saturation during the test.
  Interventions: Other: 6MWT - not accompanied

INTERVENTIONS:
Other: 6MWT - accompanied — Assessor walks behind the patient
  Arms: 6MWT - assessor walks behind the patient
Other: 6MWT - not accompanied — Assessor does not walk behind the patient
  Arms: 6MWT - assessor does not walk behind the patient

SUMMARY:
The six-minute walk test (6MWT) is a well established field exercise test to assess the functional exercise capacity in chronic obstructive pulmonary disease (COPD). The objective of this study is to assess the impact of walking behind the patient on 6MWT distance in patients with COPD.

DETAILED DESCRIPTION:
In a single-center, randomized crossover study, the investigators aim to elucidate whether there is a difference in the 6MWT distance when the assessor walks behind the patient compared to the patient walking alone.

Patients with COPD referred for pulmonary rehabilitation will be invited to perform an accompanied 6MWT (assessor walks behind the patient) and unaccompanied 6MWT (assessor does not walk behind the patient) in random order.

The tests will be performed at the end of a pulmonary rehabilitation program, after patients are familiarised with the 6MWT testing procedure and learning effects can be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of COPD according to GOLD II-IV (FEV1/FVC < 0.7, FEV1%Norm < 80%)

Exclusion Criteria:

* Inability to perform a 6MWT when arriving at the clinic (e.g., lower limb joint surgery within preceding 3 months, unstable cardiac disease, predominant neurological limitations)
* Inability to understand the instructions of the 6MWT, either of language or cognitive reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | During pulmonary rehabilitation, approximately 14 days
  Difference in six minute walk test distance between the two experimental conditions (in meter)

SECONDARY OUTCOMES:
Six minute walk test | During pulmonary rehabilitation, approximately 14 days
  Difference in patient reported perception during the two different walking tests assessed with a self-administered questionnaire. The questionnaire contains 5 questions with five response categories: 1=not at all; 2 = somewhat; 3=modestly; 4=strongly; 5= very strongly

OTHER OUTCOMES:
Oxygen saturation | During pulmonary rehabilitation, approximately 14 days
  Difference in oxygen saturation profiles between the two experimental conditions

CONTACTS AND LOCATIONS:
Overall Officials: Anja Frei, PhD, Principal Investigator — University of Zurich, EBPI, Switzerland
Locations (2):
- Switzerland (2):
  - Berner Rehazentrum AG, Heiligenschwendi, Canton of Bern
  - University of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No